CLINICAL TRIAL: NCT05702658
Title: The Effectiveness of an Autistic-delivered Peer-support Intervention for Autistic Adults: Community Autism Peer Specialist (CAPS) Program
Acronym: CAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Temple University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lindsay Shea, Associate Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206009290; 1R34MH130830 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Autism
Keywords: peer support; adult; developmental disabilities; independent living; participation
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Individuals who receive CAPS
  Interventions: Behavioral: CAPS
- control (No Intervention): Individuals who receive treatment as usual

INTERVENTIONS:
Behavioral: CAPS — Community Autism Peer Support is a one-to-one autistic-delivered peer support, community-based intervention focused on independent living and participation.
  Arms: experimental arm

SUMMARY:
The number of autistic adults reached 5.4 million in the United States in 2017 and is projected to continue to rise, but evidence-based practices to optimize their health and well-being are limited and poor outcomes are common. This study will leverage existing infrastructure to finalize the development of a novel support service provided by peers with lived experience, incorporating input from autistic peer specialists, autism researchers, peer support researchers, and experts in peer support training. Investigators will then conduct a pilot randomized controlled trial to examine the effectiveness of the service while also examining the feasibility, acceptability, and implementation procedures in preparation for future large-scale testing and dissemination.

DETAILED DESCRIPTION:
Approximately 5.4 million adults in the United States (1 in 45) are believed to have autism spectrum disorder (ASD), but there is a lack of services available to support them in reaching their full potential. Although typically conceptualized as a childhood disorder, ASD-related service needs persist into adulthood. The core social and communication impairments of ASD, reported difficulties with change, and a high rate of co-occurring mental health conditions often result in limited participation in major life areas that are determinants of health, including social and community participation, employment, housing, and transportation. The transition to adulthood is not only associated with developmental challenges, but also a "services cliff" whereby supports and services that were previously available through the education system are no longer available. Peer-delivered interventions have emerged as a potent, evidence-based modality for enhancing outcomes among other clinical populations, such as adults with serious mental illnesses, with effectiveness in enhancing social networks, empowering participants, reducing the use of inpatient services, and increasing life satisfaction. At present, there is limited research on the effectiveness of autistic-led peer support interventions, especially those that target broad aspects of community functioning. The proposed study seeks to refine, manualize, and test a pilot autistic peer support program aimed at supporting community participation among autistic young adults, with the goal of preparing it for large-scale testing and future dissemination and sustainability. The first aim of this proposal is to enhance the structure of a pilot autistic-peer delivered intervention (Community Autism Peer Specialists, or CAPS) that is currently in use as a Medicaid-reimbursed service in Philadelphia. This will include developing a manual and fidelity tool to facilitate evaluation and systematic implementation. The second and third aims are to conduct a hybrid type 1 effectiveness-implementation randomized controlled trial with 40 young autistic adults to test the feasibility and acceptability of the intervention and research procedures, while also examining proposed target mechanisms of action (e.g., self-efficacy, working alliance, perceived social support) and clinical outcomes such as community participation, loneliness, and resilience. This work will gather additional evidence and implementation information to support a fully-powered R01- funded clinical trial. The proposed efforts will involve substantial engagement of a diverse group of autistic adults in all phases along with multiple community partners, including a Medicaid payer. The project has tremendous potential to expand service options for autistic adults and is uniquely poised to have broad, scalable impact.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* Have a diagnosis of autism spectrum disorder that is confirmed by a licensed healthcare provider
* Self-reported challenges in one or more major life areas (i.e., social, school, work, self-maintenance)
* Express a desire to enhance functioning in one of these areas
* Reside in Philadelphia County
* Be able to communicate in English (i.e., understand at a basic conversational level and communicate verbally or using technology or other approaches). This is required because the intervention will be delivered in English, and the interactions between the peer specialists and participants will be in English.
* Be able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent, as assessed by research staff using an active recall method.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals will be asked to self-report their gender identity.
Enrollment: 40 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in general Self-Efficacy | Baseline, month 3, month 12
  General Self-Efficacy Scale (GSES) is a 10-item scale that will be used to measure an individual's perceptions regarding their ability to manage novel situations. All 10 items are scored using a Likert rating scale, ranging from 1 (not at all true) to 4 (exactly true).The total score ranges from 10 to 40. A higher score indicates better self-efficacy.
Change in Internalized Stigma | Baseline, month 3, month 12
  The Brief version of the Internalized Stigma of Mental Illness (ISMI-10) scale will be adapted to determine the extent to which autistic individuals have accepted perceptions from others about their ability to function successfully in the community. Each question is rated as 1= strongly disagree, 2= disagree, 3= agree, 4= strongly agree. Total scores range from 10-40, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Change in coping skills | Baseline, month 3, month 12
  The Brief COPE is a questionnaire to assess the usual coping strategies. A total of 28 items are scored on from 1=not at all to 4 = a lot, with minimum score of 28 and maximum score of 112. A higher score reflect a higher level of coping skills
Change in self-identity | Baseline, month 3, month 12
  The adapted Questionnaire on Disability Identity and Opportunity (QDIO) uses 30 questions to measure disability participation and orientation, using a five-point Likert scale where 1 = strongly disagree and 5 = strongly agree. Total scores range from 30 to 150, with higher score reflecting a more positive self-identity
Change in social support | Baseline, month 3, month 12
  The Patient-Reported Outcomes Measurement Information System (PROMIS) emotional support and informational support item banks will be used to measure social support. A total of 8 items are scored on a 5-point response scale. Scores can range from 8 to 40 (a higher score means higher reported support).
Change in unmet needs | Baseline, month 3, month 12
  A modified version of the Camberwell Assessment of Need will be used to assess unmet needs in 23 life domains, including housing, taking care of one's home, autism information and treatment, psychological distress, social life, intimate relationships, and other areas. The total scores range from 0 to 23, with higher score indicating more unmet needs
Change in social functioning | Baseline, month 3, month 12
  The Social Responsiveness Scale, 2nd edition (SRS-2) is among the most well-validated and frequently used measures of ASD symptomatology. The SRS-2 provides a continuous measure of social ability. Scores range from 30 to >= 90, with higher scores indicating greater social impairment.
Change in Cognitive Flexibility | Baseline, month 3, month 12
  The Shift scale from the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) will be used to measure cognitive flexibility. Participants rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience within the last month. The sum of 6 items yields the raw score (range: 6-18). A lower score represents a better outcome.
Change in Loneliness | Baseline, month 3, month 12
  The University of California Los Angeles Loneliness Scale, Version 3 is a 20-item scale that assesses feelings of loneliness and social isolation. Participants rate items on a 4-point Likert scale ranging from 1 (never) to 4 (often).Items are summed to create a score that can range from 20-80, higher scores being indicative of greater loneliness.
Change in Purpose in Life | Baseline, month 3, month 12
  The PROMIS Meaning and Purpose item bank that consists of 8 items will be used. The response options range from "not at all" to "very much," yielding a raw score from 8 to 40. A higher score indicates a higher level of purpose in life.
Change in Resilience | Baseline, month 3, month 12
  The Connor-Davidson Resilience Scale - 10 (CD-RISC) is the most frequently used instrument to measure resilience. The measure consists of 10 items using a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all of the time). The scale measures how the participant felt over the past month. The questionnaire produces an overall resilience score that ranges from 0-40, with higher scores representing greater resilience.
Change in Hope | Baseline, month 3, month 12
  The Adult Hope Scale assesses belief in one's own ability to pursue desired goals and employ strategies needed to achieve the goals. A total of 12 items are scored on a scale from 1=Definitely False to 8 =Definitely True. Total scores range from 12 to 96, with a higher score reflecting a higher level of perceived hope.
Changes in Community Participation | Baseline, month 12
  We will use a modified version of the Temple University Community Participation Measure (TUCP) to measure community participation. A total of 27 items measure the total days of participation (ranging from 0 - 810) and total participation areas (ranging from 0-27), with higher scores indicating higher levels of community participation.
Changes in Quality of Life | Baseline, month 12
  WHOQOL-BREF evaluates both objective and subjective aspects of quality of life. A total 26 item produces four domain scores: physical, psychological, social relationships and environment domain (Likert type scale ranging from 1- strongly disagree to 5 - strongly agree). The total scores range from 26 to 130, with a higher score reflecting a higher level of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the NIMH Data Archive